CLINICAL TRIAL: NCT02357823
Title: Long Term Serological Response and Memory Cells Role After Different Pneumococcal Vaccine Strategies in HIV Adults
Brief Title: Antibodies and Memory Cells Role After Different Pneumococcal Vaccines in HIV Adults
Status: Withdrawn | Type: Observational
Sponsor: University of Siena (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesca Montagnani, Md, PhD, University of Siena
Other Study IDs: PCV13HIV-BOOST-2013
Record Dates: First submitted 2015-01-22; First posted 2015-02-06 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: HIV; Pneumococcal Infections
Keywords: Pneumococcal vaccine; HIV infection; 13-valent Pneumococcal Conjugate Vaccine; 23-valent Pneumococcal Polysaccharide Vaccine
MeSH Terms: conditions — Pneumococcal Infections; HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbes isolated from nasopharingeal swab; blood for analysis of immune response
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group 1: Immunological and microbiological status of HIV- positive adults with pneumococcal vaccinal status of 2 PCV13 doses received from more than 3 years that have prescription for a single booster dose of PCV13.
  Interventions: Other: Evaluation of immunological response; Other: Nasopharyngeal swabs analysis
- Group 2: Immunological and microbiological status of HIV- positive adults with pneumococcal vaccinal status of 1 PPV23 dose received from more than 3 years that have prescription to receive 2 doses (priming + boost) of PCV13.
  Interventions: Other: Evaluation of immunological response; Other: Nasopharyngeal swabs analysis
- Group 3: HIV- positive adults that have never received a pneumococcal vaccine (naive) and have a CD4+ cell count < 200 cells/ul that have prescription to be primed with a single dose of PCV13 then boosted with a single dose of PPV23.
  Interventions: Other: Evaluation of immunological response; Other: Nasopharyngeal swabs analysis
- Group 4: Immunological and microbiological status of HIV- positive adults that have never received a pneumococcal vaccine (naive) and have a CD4+ cell count > 200 cells/ul that have prescription to be primed with a single dose of PCV13 then boosted with a single dose of PPV23.
  Interventions: Other: Evaluation of immunological response; Other: Nasopharyngeal swabs analysis
- Group 5: Immunological and microbiological status of HIV- positive adults with pneumococcal vaccinal status of 1 PPV23 dose received from more than 3 years and that that have prescription to receive a single dose of PCV13.
  Interventions: Other: Evaluation of immunological response; Other: Nasopharyngeal swabs analysis

INTERVENTIONS:
Other: Evaluation of immunological response — Study of short and long term immunological response after different schedule of PCV13 or PPV23
Other: Nasopharyngeal swabs analysis — Evaluation of pneumococcal nasopharyngeal colonization

SUMMARY:
Streptococcus pneumoniae is a cause of high morbidity and mortality in HIV-positive subjects, representing the leading etiological agent of severe bacterial pneumonia. International guidelines recommend that HIV positive patients aged >=19 years, who are 13-valent conjugate vaccine (PCV13) naïve, should receive a single dose of PCV13. Pneumococcal polysaccharide vaccine 23-valent (PPV23) should be given >=8 weeks after indicated dose of PCV13, and a second dose of PPV23 should be given 5 years later. For those who previously received PPV23, PCV13 should be administered >=1 year after the last PPV23 dose. HIV infection affects humoral immunity both through reduced T-cell help and changes in the B-cell compartment. Neither amount of circulating memory B cells nor their functions are restored by antiretroviral therapy: this may affect antibody mediated immunity, even in well-treated HIV patients. In asplenic childrens a single dose of PCV13 seems sufficient to restore the pool of anti-pneumococcal polysaccharides IgG memory B cells. In adults, it has been reported that a single dose of 7-valent pneumococcal conjugate vaccine induces significant increases in serotype-specific memory B-cell populations, conversely, immunization with PPV23 seems to decrease memory B-cell frequency. However, data on immunological response after PCV13 in HIV positive adults are still scanty and the optimal pneumococcal prophylaxis strategy needs further investigation. Number of PCV13 doses is actually demanded to clinical judgment for each patient; also current Italian indications recommend at least one dose, but till 3 doses seem to be suggested for immunocompromised patients. Present study aims to investigate short and long term immunological response after different standard vaccine schedule and to evaluate pneumococcal nasopharyngeal colonization in vaccinated patients.

DETAILED DESCRIPTION:
The study will be divided in 3 main aims; in the first, the long term immunological response to PCV13 and PPV23 in HIV+ adults will be evaluated. In a previous clinical trial (PRIN 2009 study, Clinicaltrials: NCT02123433) a cohort of HIV positive adults had been vaccinated either with 2 doses of PCV13 8 weeks apart or 1 dose of PPV23 (last enrollment: December 2012). Immunoglobulins G (IgGs) against 12 common pneumococcal serotypes included in PCV13 and PPV23 were quantified by ELISA at baseline (BL), 8, 24 and 48 weeks: analysis are still ongoing; preliminary data revealed that both vaccines were safe and well tolerated and showed similar immunogenicity. The present study aims to evaluate persistence of long term (>= 3 years) serological and memory B cells response in those previous vaccinated groups. In this phase, population will be screened for inclusion and exclusion criteria to entire study conduction. Once obtained informed consent, patients will be enrolled. Together with the collection of blood samples for routine purposes, an additional blood sample will be taken so to run immunological tests (ELISA, ELISpot). It is important to underline that no invasive procedures are needed for the study, apart from routine clinical practice: blood specimens will be obtained as part of routine investigations, blood will be hence taken for CD4+ cell count, viraemia analysis and anti-HIV drug monitoring; enrolled patients will agree just to donate a blood sample for research purposes. Blood samples will be collected from all previously PCV13 or PPV23 vaccinated HIV+ subjects and serum antibodies and B cells isotypes will be analyzed at baseline (BL), that is >= 3 years after a previous PCV13 or PPV23 vaccination.

The second objective of this study aims to evaluate short and long term immunological response with different combined vaccine strategies in HIV+ adults. Participants will be recruited if they'll have needed to receive antipneumococcal vaccines (primary or booster) according to clinical standard indications.

Elicited immunological response (serum antibodies and B cells isotypes) will be explored at BL, 8, 24, 48 and 96 weeks after additional different received pneumococcal vaccine strategies. At BL, after collecting blood samples as previously described for Aim1, every patient will be assigned to a specific Group on the basis of the received vaccine schedule, prescribed by clinicians according to individual clinical indications. Short- (30 minutes), medium- (<=5 days) and long-term adverse reactions will be reported, by clinical evaluation within 30 minute post-vaccine, phone call at day 5 and anamnestic data collection during follow up 8, 24, 48 and 96 weeks.

Blood samples will be analyzed at 8, 24, 48 and 96 weeks to evaluate serum antibodies and B cells isotypes.

Finally, the third aim of the study will lead an epidemiological and microbiological survey in vaccinated HIV+ adults. At BL, 8, 24, 48 and 96 weeks all clinical-anamnestic data will be updated, together with blood sample analysis to title IgG towards each vaccinal pneumococcal polysaccharides and to evaluate B cells isotypes and nasopharyngeal swab for S. pneumoniae culture, in vitro chemosusceptibility tests, serotyping, clonal analysis by Multilocus Locus Sequence Typing (MLST).

Carriage will be defined as S. pneumoniae isolation from one or more of the nasal swabs, in absence of any clinical signs or symptoms; a 12 months clinical follow up will be performed in colonized patients. All patients developing infections will be followed until resolution.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* acceptance of informed consensus
* HIV positivity
* access to structures in ambulatory or Day Hospital regimen
* CD4+ cell count > or < than 200 cells/ul
* subjects for which Italian Ministry of Health recommend pneumococcal vaccination with PCV13 or PPV23

Exclusion Criteria:

* pregnancy
* acute infectious disease ongoing
* antibiotic therapy ongoing in the previous 7 days
* HIV-independent immunodepression
* chronic steroid therapy
* anatomic or functional asplenia
* contraindication to vaccination based on package insert drug facts, such as hypersensitivity to the active ingredient or one of the bulking agents (PPV23, Pneumovax);hypersensitivity to the active ingredient, to one of the bulking agents or to the diphteria toxoid (PCV13, Prevenar 13)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-positive adults that undergo the International and Italian Ministry of Health indications for administration of pneumococcal vaccines.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Immunological response evaluation | 24 months
  Dosing of serotype specific antibodies (cut off value: 0.35 mcg/mL for each vaccine polysaccharide antigen) and quantification of number and phenotype of serotype specific B cells

SECONDARY OUTCOMES:
Streptococcus pneumoniae colonization | 24 months
  Presence of S. pneumoniae in nasopharyngeal swabs culture

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Montagnani, MD, PhD, Principal Investigator — Università degli Studi di Siena - Dipartimento di Biotecnologie Mediche - Dipartimento di Malattie Infettive Universitarie
Locations (2):
- Italy (2):
  - Istituto di Clinica delle Malattie Infettive c/o Policlinico Gemelli, Largo Agostino Gemelli 12, Roma, Rome
  - UOC Malattie Infettive Universitarie c/o Policlinico Le Scotte, Viale Mario Bracci 16, Siena

REFERENCES:
- [Result] Rubin LG, Levin MJ, Ljungman P, Davies EG, Avery R, Tomblyn M, Bousvaros A, Dhanireddy S, Sung L, Keyserling H, Kang I; Infectious Diseases Society of America. 2013 IDSA clinical practice guideline for vaccination of the immunocompromised host. Clin Infect Dis. 2014 Feb;58(3):309-18. doi: 10.1093/cid/cit816. PMID 24421306
- [Result] Clutterbuck EA, Lazarus R, Yu LM, Bowman J, Bateman EA, Diggle L, Angus B, Peto TE, Beverley PC, Mant D, Pollard AJ. Pneumococcal conjugate and plain polysaccharide vaccines have divergent effects on antigen-specific B cells. J Infect Dis. 2012 May 1;205(9):1408-16. doi: 10.1093/infdis/jis212. Epub 2012 Mar 29. PMID 22457293
- [Result] Lu CL, Hung CC, Chuang YC, Liu WC, Su CT, Hsiao CF, Tseng YT, Su YC, Chang SF, Chang SY, Chang SC. Comparison of serologic responses to vaccination with one dose or two doses of 7-valent pneumococcal conjugate vaccine in HIV-infected adult patients. Vaccine. 2012 May 21;30(24):3526-33. doi: 10.1016/j.vaccine.2012.03.070. Epub 2012 Apr 4. PMID 22484349
- [Result] Klugman KP, Madhi SA, Feldman C. HIV and pneumococcal disease. Curr Opin Infect Dis. 2007 Feb;20(1):11-5. doi: 10.1097/QCO.0b013e328012c5f1. PMID 17197876